CLINICAL TRIAL: NCT05606666
Title: Reliability of the Neurophysiology of Pain Questionnaire in the Neck Pain the Cross-validation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Özden Laçin, MsC, Istanbul Arel University
Other Study IDs: NPQ Cross-validation
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Neck Pain; Pain Knowledge
Keywords: neck pain; neurophysiology of pain; pain knowledge; pain education
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: reliability of the NPQ — The aim of this study is to study the validity and reliability of the Modified Pain Neurophysiology Questionnaire in patients with neck pain.

SUMMARY:
The aim of this study is to study the validity and reliability of the Modified Pain Neurophysiology Questionnaire in patients with neck pain. After the ethics committee approval, women and men in Turkey will be invited to the research via online advertisements (researchers' facebook, instagram, twitter accounts). The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained with a common opinion from these two Turkish translations. In ten trial phases, a preliminary assessment will be conducted with 15 participants to test the intelligibility of the scale. If there are participants who think that there is a problem with the intelligibility of the scale, they will be asked to explain which items they have problems understanding and why. After individuals are informed with the online voluntary consent form, participants will be asked to complete the Modified Pain Neurophysiology questionnaire. Modified Pain Neurophysiology scale questions and questions in the data collection form will be prepared through the google surveys application and will be sent to the participants via Whatsapp, Facebook, Instagram and e-mail. Participants will fill out the survey forms online. In order to evaluate the validity of the Modified Pain Neurophysiology questionnaire, the pain subscale of the SF-36 scale, which has been validated in Turkish, will be used (McHorney, Ware, Lu, and Sherbourne, 1994), (Kocyigit et al., 1999). Scales after 15 days to assess test-retest reliability will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-65
* Having neck pain complaints for the last 3 months
* Adult individuals who agreed to participate in the study. Their mother tongue is Turkish.

Exclusion Criteria:

* Not answering all the questions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons who meet the inclusion criteria and who volunteered to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
pain subscale of the SF-36 questionnaire | baseline
  We will use only the pain subscale of the validated Turkish version of the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul, Istanbul, Turkey (Türkiye)